CLINICAL TRIAL: NCT04024332
Title: A Single-center, Open-label, Single-dose Study to Investigate the Pharmacokinetics of ACT-541468 in Subjects With Severe Renal Impairment Compared to Healthy Subjects
Brief Title: Study of the Way the Body Takes up, Distributes, and Gets Rid of ACT-541468 in Subjects With Abnormal Kidney Function Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID-078-115; 2019-002159-40 (EudraCT Number)
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Renal Insufficiency; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, single-dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (healthy) (Experimental): On Day 1, 8 healthy subjects will receive a single oral dose of 25 mg ACT-541468 in fasted condition.
  Interventions: Drug: ACT-541468
- Group B (severe renal function impairment) (Experimental): On Day 1, 8 subjects with severe renal function impairment will receive a single oral dose of 25 mg ACT-541468 in fasted condition.
  Interventions: Drug: ACT-541468

INTERVENTIONS:
Drug: ACT-541468 — ACT-541468 25 mg; administered orally

SUMMARY:
Study of the way the body takes up, distributes, and gets rid of ACT-541468 in subjects with abnormal kidney function compared to healthy subjects

ELIGIBILITY:
General inclusion criteria for all subjects:

* Signed informed consent in the local language prior to any study mandated procedure.
* Male and female subjects aged 18 to 85 years (inclusive) at screening.
* Body mass index (BMI) from 18 to 35 kg/m2 (inclusive) at screening. Body weight at least 50 kg.
* Women of childbearing potential: Women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use (during the entire study and 30 days thereafter) a highly effective method of contraception with a failure rate of < 1% per year.
* Women of non-childbearing potential, i.e., postmenopausal, XY genotype, Turner syndrome, uterine agenesis: no contraceptive requirement.

Additional inclusion criteria for healthy subjects (Group A):

* Normal renal function as confirmed based on Creatinine Clearance (CLcr) by the Cockcroft-Gault equation adjusted for age: >= 80 mL/min for subjects <= 50 years of age; >= 70 mL/min for subjects 51-60 years of age; >= 60 mL/min for subjects 61-85 years of age; CLcr = ([140-age(years)]×weight (kg))/(72×serum creatinine (mg/dL)) (x 0.85 for female subjects)
* The CLcr value should be confirmed (± 25%) on Day -1 in case subjects will be dosed more than 10 days after the day of screening.
* Hematology, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening.
* Each healthy subject must be matched with one subject with severe renal function impairment with regard to age (± 10 years difference allowed), body weight (± 15% difference allowed), and sex, determined by results at screening.

Additional inclusion criteria for subjects with severe renal function impairment (Group B)

* Severe renal function impairment as confirmed based on CLcr by the Cockcroft-Gault equation: <30 mL/min, not on dialysis.
* The CLcr value should be confirmed (± 25%) on Day -1 since subjects will be dosed more than 10 days after the day of screening.
* Hematology, clinical chemistry, coagulation and urinalysis test results consistent with severe renal function impairment at screening.
* Physical examination without clinically relevant abnormalities at screening and on Day -1 (except for those related to severe renal function impairment), which would interfere with the objectives of the study.
* Stable concomitant medications.

General exclusion criteria for all subjects:

* Pregnant or lactating women.
* Clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal
* History of renal and/or liver transplant.
* Hepatic cancer, primary biliary cirrhosis or any form of cholestatic disease.
* Use of drugs which might interfere with the PK of ACT-541468 (moderate to strong CYP3A4 inhibitors or inducers).
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Additional exclusion criteria for healthy subjects (Group A)

* History or clinical evidence of any unstable disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study treatment (appendectomy, herniotomy, and cholecystectomy allowed).
* Intake of any creatine supplement from screening to EOS.

Additional exclusion criteria for subjects with severe renal function impairment (Group B).

- End-stage renal disease that requires dialysis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
AUC of ACT-541468 from time zero to 24 h after study drug administration (AUC0-inf) | Blood samples for PK analysis will be taken at multiple time points after ACT-541468 administration for a total duration of up to 4 days

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent (serious) adverse events (S)AEs | During treatment with ACT-541468 administration for a total duration of up to 4 days

OTHER OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-541468 | Blood samples for PK analysis will be taken at multiple time points after ACT-541468 administration for a total duration of up to 4 days
Time to reach maximum plasma concentration (tmax) of ACT-541468 | Blood samples for PK analysis will be taken at multiple time points after ACT-541468 administration for a total duration of up to 4 days
Terminal half-life (t½) of ACT-541468 | Blood samples for PK analysis will be taken at multiple time points after ACT-541468 administration for a total duration of up to 4 days
Extent of plasma protein binding (PPB; in %) | Blood samples for PK analysis will be taken at multiple time points after ACT-541468 administration for a total duration of up to 4 days
  PPB % = 100 - (Cu/C×100), with 'Cu' standing for unbound and 'C' for total plasma ACT-541468 concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- APEX GmbH, München, Germany

IPD SHARING:
Plan to Share IPD: No